CLINICAL TRIAL: NCT01537900
Title: A Multiple Dose Study to Evaluate Pharmacokinetics and Hepatitis C Virus RNA Dynamics Following Administration of MK-5172 in Hepatitis C Infected Patients
Brief Title: A Multiple Dose Study of Grazoprevir (MK-5172) in Hepatitis C-Infected Participants (MK-5172-010)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5172-010; 2011-000435-83 (EudraCT Number)
Record Dates: First submitted 2012-02-17; First posted 2012-02-23 (Estimated); Results first posted 2016-03-04 (Estimated); Last update posted 2018-09-14 (Actual); Status verified 2018-08

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — grazoprevir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Grazoprevir 100 mg (Experimental): Participants received GZR 100 mg once daily (q.d.) for 7 days. Liver FNA was performed on Day 7.
  Interventions: Drug: Grazoprevir

INTERVENTIONS:
Drug: Grazoprevir — GZR 100 mg tablet by mouth q.d. for 7 days.
  Other Names: MK-5172

SUMMARY:
The goal of this study was to compare hepatic pharmacokinetics (PK) derived from liver tissue to plasma PK after administration of grazoprevir (MK-5172) to participants with chronic hepatitis C virus (HCV) infection. Participants will be randomized to one of four different liver ultrasound-guided Fine Needle Aspirate (FNA) schedules (at 4-, 8-, 24-, or 72-hours after the Day 7 dose).

ELIGIBILITY:
Inclusion criteria:

* has a Body Mass Index (BMI) ≥18.5 kg/m² and ≤36.0 kg/m²
* has chronic compensated, genotype 1 HCV infection
* has no cirrhosis of the liver as confirmed by FibroSure®/Fibro Test® and/or local country procedure (e.g. transient elastography/Fibroscan)
* does not require anticoagulants, nonsteroidal anti-inflammatory agents, and aspirin for at least fourteen (14) days preceding the initial liver biopsy and continuing throughout the entire study
* if is a female participant of reproductive potential, is willing to use 2 medically acceptable forms of contraception for 2 weeks prior to start of treatment through 2 weeks after last study treatment
* if is a male participant with a partner(s) of reproductive potential, is willing to use 2 medically acceptable forms of contraception from first dose to 90 days after last dose

Exclusion criteria:

* has a history of stroke, chronic seizures, or major neurological disorder
* has received previous treatment with a direct-acting antiviral (DAA)
* has evidence of high grade bridging fibrosis from prior liver biopsy within 3 years of study entry
* has evidence or history of chronic hepatitis not caused by HCV infection including but not limited to non-HCV viral hepatitis, nonalcoholic steatohepatitis (NASH), drug-induced hepatitis, or autoimmune hepatitis
* has clinical or laboratory evidence of cirrhosis or other advanced liver disease
* has decompensated liver disease as indicated by a history of ascites, hepatic encephalopathy, or bleeding esophageal varices
* has been diagnosed with, or suspected of having, hepatocellular carcinoma (HCC)
* has clinically significant abnormality on an electrocardiogram (ECG)
* is co-infected with human immunodeficiency virus (HIV)
* is positive for Hepatitis B surface antigen (HBsAg) or other evidence of active Hepatitis B infection
* has a history of gastric bypass surgery, bowel resection or other disorder that may interfere with absorption
* has a history of clinically significant uncontrolled endocrine, gastrointestinal, cardiovascular, hematological, immunological, renal, respiratory, or genitourinary abnormalities or diseases
* has clinically significant neoplastic disease
* uses alcohol to excess, defined as greater than 3 glasses of alcoholic beverages (1 glass is approximately equivalent to: beer [354 mL], wine [118 mL], or distilled spirits [29.5 mL]) per day
* is a current regular user (including use of any illicit drugs) or history of drug (including alcohol) abuse within the last 3 months
* has undergone surgery, donation of 1 unit of blood (approximately 500 mL) or participation in another investigational study within a period of 4 weeks prior to the screening visit
* has a history of multiple and/or severe allergies, or anaphylactic reaction or intolerability to prescription or nonprescription drugs or food
* is pregnant or lactating
* is expecting to donate eggs or sperm

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2014-07-31 (Actual); Study Completion 2014-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Grazoprevir 100 mg
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Grazoprevir 100 mg: Participants received GZR 100 mg q.d. for 7 days. Liver FNA was performed on Day 7.
Arm/Group | Grazoprevir 100 mg
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.5 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Estimated Area Under the Liver Concentration-time Curve for 24 Hours Post-dose (AUC[H]0-24hr) of Grazoprevir
Description: Each participant was assigned to undergo Fine Needle Aspiration (FNA) to obtain liver tissue at different time points. Specifically, one participant underwent FNA at 4 hr post-dose only, another participant underwent FNA at 8 hr post-dose only, and a third participant underwent FNA at 24 hr post-dose only. (The fourth participant underwent FNA at 72 hr post-dose and therefore was not included in the calculation of AUC0-24hr.) Therefore, in calculating AUC0-24hr, there were only 3 data points: 1 data point at 4 hr post-dose, 1 data point at 8 hr post-dose, and 1 data point at 24 hr post-dose. The model assumed that drug concentration was at steady-state, and that the concentration at 24 hr post-dose was equal to the concentration at 0 hr post-dose.
Time Frame: 4, 8, and 24 hours post-dose on Day 7
Population: The per protocol population (PPP) includes all participants (4, 8, and 24 hr time points) who complied with the protocol sufficiently to ensure that the data were likely to exhibit the effects of treatment. As each data point was obtained from unique participants, there is no measure of variability.
Measure: Number; unit: µM*hr
Arm/Group | Grazoprevir 100 mg
Number analyzed (Participants) | 3
µM*hr | 19800

2. Primary Outcome: Hepatic Concentration of GZR (C[H]Xhr)
Description: C(H)Xhr of GZR was expressed as liver concentration (μmol GZR/L liver) using the concentration of the extracted liver sample (mass of the liver biopsy/0.2 mL solvent), and assuming that liver has the specific gravity of water (1 g/mL). The arithmetic mean C(H)Xhr concentration is based on the means of 4 FNA passes per participant in all 4 participants.
Time Frame: 4, 8, 24, and 72 hours post-dose on Day 7
Population: The PPP includes all participants who complied with the protocol sufficiently to ensure that the data were likely to exhibit the effects of treatment.
Measure: Mean (Standard Deviation); unit: µM
Arm/Group | Grazoprevir 100 mg
Number analyzed (Participants) | 4
µM
  Hepatic concentration at 4 hours (C[H]4hr) | 390 (186)
  Hepatic concentration at 8 hours (C[H]8hr) | 1340 (1335)
  Hepatic concentration at 24 hours (C[H]24hr) | 575 (505)
  Hepatic concentration at 72 hours (C[H]72hr) | 434 (108)

3. Primary Outcome: Apparent Terminal Hepatic Half-life (t[H]½ ) of GZR
Description: t(H)1/2 is a measure of the time required for the maximum post-dose liver concentration of GZR to decrease by 50%.
Time Frame: 4, 8, 24, and 72 hours post-dose on Day 7
Population: Apparent t(h)1/2 could not be estimated due to insufficient data in the terminal phase.
Arm/Group | Grazoprevir 100 mg
Number analyzed (Participants) | 0

4. Secondary Outcome: Plasma AUC[0-24 hr] of GZR
Description: AUC0-24hr is a measure of the mean concentration of drug in plasma after dosing to 24 hours post-dose.
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 48 and 72 hours post-dose on Day 7
Population: Plasma PK data were not collected due to liver PK results being deemed physiologically impossible.
Arm/Group | Grazoprevir 100 mg
Number analyzed (Participants) | 0

5. Secondary Outcome: Maximum Plasma Concentration (Cmax) of GZR
Description: Cmax is a measure of the maximum plasma concentration post-dose.
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 48 and 72 hours post-dose on Day 7
Population: Plasma PK data were not collected due to liver PK results being deemed physiologically impossible.
Arm/Group | Grazoprevir 100 mg
Number analyzed (Participants) | 0

6. Secondary Outcome: Lowest Plasma Concentration (Ctrough) of GZR
Description: Ctrough is a measure of drug concentration 24 hours post-dose.
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 48 and 72 hours post-dose on Day 7
Population: Plasma PK data were not collected due to liver PK results being deemed physiologically impossible.
Arm/Group | Grazoprevir 100 mg
Number analyzed (Participants) | 0

7. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of GZR
Description: Tmax is a measure of time to reach maximum post-dose plasma drug concentration.
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 48 and 72 hours post-dose on Day 7
Population: Plasma PK data were not collected due to liver PK results being deemed physiologically impossible.
Arm/Group | Grazoprevir 100 mg
Number analyzed (Participants) | 0

8. Secondary Outcome: Plasma t½ of GZR
Description: t1/2 is a measure of time for the maximum plasma concentration of GZR to decrease by 50%.
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 48 and 72 hours post-dose on Day 7
Population: Plasma PK data were not collected due to liver PK results being deemed physiologically impossible.
Arm/Group | Grazoprevir 100 mg
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From Screening up to 14 days after final dose (up to Day 21)
Arm/Group | Grazoprevir 100 mg
Serious Adverse Events (participants affected / at risk) | 1/4
Other Adverse Events (participants affected / at risk) | 1/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Grazoprevir 100 mg (N=4)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Grazoprevir 100 mg (N=4)
Diarrhoea (Gastrointestinal disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation.